CLINICAL TRIAL: NCT01318811
Title: A Comparison of Dilute Unfractionated Heparin and Standard Concentrated Unfractionated Heparin Protocols for Anticoagulation of the Extra-corporeal Circuit During Continuous Renal Replacement Therapy in the ICU
Brief Title: A Comparison of Dilute Versus Concentrated Heparin for CRRT Anticoagulation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Thomas Golper, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VU 110162
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury; Acute Renal Failure; Heart Failure
Keywords: Heparin; CRRT; Continuous renal replacement therapy; CVVHD; Anticoagulation
MeSH Terms: conditions — Acute Kidney Injury; Heart Failure | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dilute heparin (Active Comparator): Arm A will receive dilute heparin delivered as an intravenous infusion proximal to the dialysis filter.
  Interventions: Drug: Dilute unfractionated heparin
- Standard concentrated heparin (Active Comparator): Arm B will receive standard concentrated heparin and will be delivered as an intravenous infusion proximal to the dialysis filter.
  Interventions: Drug: Standard concentration unfractionated heparin

INTERVENTIONS:
Drug: Dilute unfractionated heparin — Patients in the dilute heparin arm will receive a systemic loading dose of heparin of 15 units per kilogram of weight by rapid intravenous bolus. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started. Heparin will be delivered as a solution of 2 units/mL and the infusion will be prepared with 2,000 units of heparin in 1,000 mL of 0.9% NaCl and delivered intravenously proximal to the dialysis filter.
  Other Names: Heparin
  Arms: Dilute heparin
Drug: Standard concentration unfractionated heparin — Patients in the standard heparin arm will receive a systemic loading dose of heparin of 15 units per kilogram of weight by rapid intravenous bolus. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started and delivered in a standard concentration intravenously proximal to the dialysis filter via a syringe. The concentration of heparin used will be 1,000 units of heparin per 1 mL of 0.9% NaCl.
  Other Names: Heparin
  Arms: Standard concentrated heparin

SUMMARY:
Heparin is commonly used for anticoagulation of the extracorporeal circuit during continuous renal replacement therapy (CRRT) but the optimal mode of delivery has not yet been validated. Our study will compare dilute heparin to a standard concentration of heparin. The investigators hypothesize that heparin delivered in a dilute solution will augment coating of the filter fibers with anticoagulants, decreasing clotting events and increasing filter life. By improving delivery of heparin to the filter and circuit, where clotting events can disrupt dialysis, less heparin would be required for the extra-corporeal circuit and thus less heparin would be delivered back to the patient with blood return from the machine. By exposing the patient to less heparin it is hypothesized that fewer bleeding events would occur, making the dialysis treatment safer. If more of the filter's fibers remain patent and the filter is functional for a longer period of time, the CRRT would also be more effective.

DETAILED DESCRIPTION:
Our study will compare two protocols using heparin for anticoagulation of the extra-corporeal circuit during CRRT. Study subjects will be recruited from patients started on continuous venovenous hemodialysis (CVVHD) in all intensive care units at Vanderbilt University Medical Center (VUMC). Once enrolled, patients will be pragmatic cluster-randomized (by month of entry) into one of two study arms. Arm A will receive dilute heparin and arm B will receive standard concentrated heparin as both approaches are standard practices at VUMC. Heparin will be delivered as an intravenous infusion proximal to the dialysis filter in both groups. Replacement of the extra-corporeal circuit, including the dialysis filter, is performed under several circumstances: stopping of CRRT when the subject is transported out of the ICU for a procedure or study, machine malfunction, and clotting of the filter. All CRRT circuits and filters, regardless of patency, are replaced at 72 hours per our dialysis unit protocol. Only data from the first filter used for CVVHD will be used and the study subject's enrollment will end with replacement of the extracorporeal circuit and filter.

Study subjects will receive standard care for the duration of the study and the inpatient Nephrology team will control all aspects of the dialysis treatment. Changes to the heparin infusion rates will be made based on the heparin nomogram for this study and it applies to either arm. A copy of this nomogram will be provided to the inpatient Nephrology team who will make adjustments to the heparin infusion as required to maintain blood anticoagulation levels at goal. The principle investigators (PIs) will be available at all times by pager and phone to address questions regarding proper adjustment of the heparin infusion and will monitor each heparin dosing change to ensure consistency in implementation of the study protocol.

The following is a summary for the two interventions (arms):

Treatment Algorithm Dilute heparin: Patients in the dilute heparin arm (enrolled in odd calendar months) will receive a systemic loading dose of heparin of 15 units per kilogram of weight (all heparin doses will be rounded to the nearest 100 units) by rapid (< 10 seconds) intravenous bolus. The heparin concentration for the rapid intravenous loading bolus is 1000 units per mL. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started. Heparin will be delivered as a solution of 2 units/mL and the infusion will be prepared with 2,000 units of heparin in 1,000 mL of 0.9% NaCl and delivered intravenously proximal to the dialysis filter.

Standard concentrated heparin: Patients in the concentrated heparin arm (enrolled in even calendar months) will receive a systemic loading dose of heparin of 15 units per kilogram of weight* by rapid (< 10 seconds) intravenous bolus. The heparin concentration for the rapid intravenous loading bolus for this arm is also 1000 units per mL. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started and delivered via a syringe on the Prismaflex® proximal to the dialysis filter. The concentration of heparin used will be 1,000 units of heparin per mL of 0.9% NaCl.

Dose monitoring and adjustment: aPTT tests will be measured at baseline and at regular intervals thereafter. Adjustment of the heparin dose will be made using a heparin nomogram (see below) if the aPTT is not at the target level of greater than 35 seconds and less than 50 seconds. aPTT levels will be monitored every six hours routinely. If a significant change is made to the heparin infusion rate due to a prolonged aPTT, the aPTT will be checked at a shorter interval of three hours to ensure that aPTT is not persistently at a supratherapeutic level as this could increase risk for bleeding complications.

Nomogram for heparin infusion:

aPTT (in seconds)< 35, infusion (continue), infusion rate change (increase 10%), repeat aPTT (in 6 hours);

aPTT (in seconds) 35 to 50, infusion (continue), infusion rate change (no change), repeat aPTT (in 6 hours);

aPTT (in seconds) 51 to 60, infusion (stop for 1/2 hour), infusion rate change (decrease 10%), repeat aPTT (in 3 hours);

aPTT (in seconds) 61 to 70, infusion (stop for 1 hour), infusion rate change (decrease 20%), repeat aPTT (in 3 hours);

aPTT (in seconds) 71 to 80, infusion (stop for 1.5 hours), infusion rate change (decrease 20%), repeat aPTT (in 3 hours);

aPTT (in seconds) >80, infusion (stop for 2 hours), infusion rate change (decrease 20%), repeat aPTT (in 3 hours);

For the purposes of this study, data will only be collected from the first filter used during the CVVHD treatment. Following the end of the study enrollment period patients will continue on CVVHD and heparin infusions at the discretion of their treating physicians. Heparin infusions will continue to be adjusted based on the heparin nomogram.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Renal failure, electrolyte disturbance, or volume overload requiring continuous venovenous hemodialysis (CVVHD) as determined by the Nephrology consult service

Exclusion Criteria:

* Age less than 18 years
* Active bleeding
* Coagulopathy as defined by baseline INR > 1.8, aPTT > 45 seconds, or platelet count < 50 thousand/μL
* Active administration of systemic anticoagulation (such as warfarin, therapeutic unfractionated heparin, or therapeutic enoxaparin)
* Contraindication to heparin (allergy, thrombocytopenia with platelet count < 50, known or suspected heparin induced thrombocytopenia [HIT])
* Contraindication to systemic anticoagulation (recent surgical or other invasive procedure, significant bleeding disorder, concern for intracranial bleeding, or other contraindication as determined by treating physician)
* Administration of drotrecogin (Xigris™)
* Anticipated surgical or other invasive procedure that would necessitate withdrawal of anticoagulation within 72 hours
* Expected termination of continuous renal replacement therapy (CRRT) or death in < 24 hours
* The need for more than 500 cc an hour of IV fluids delivered proximal to the filter for the purpose of performing continuous venovenous hemofiltration (CVVH) or continuous venovenous hemodiafiltration (CVVHDF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2016-04-03 (Actual); Study Completion 2016-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Golper, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Tolwani AJ, Wille KM. Anticoagulation for continuous renal replacement therapy. Semin Dial. 2009 Mar-Apr;22(2):141-5. doi: 10.1111/j.1525-139X.2008.00545.x. PMID 19426417
- [Background] van de Wetering J, Westendorp RG, van der Hoeven JG, Stolk B, Feuth JD, Chang PC. Heparin use in continuous renal replacement procedures: the struggle between filter coagulation and patient hemorrhage. J Am Soc Nephrol. 1996 Jan;7(1):145-50. doi: 10.1681/ASN.V71145. PMID 8808122
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078

RESULTS

PARTICIPANT FLOW:
Groups:
- Dilute Heparin: Arm B will receive dilute heparin delivered as an intravenous infusion proximal to the dialysis filter.
  Dilute unfractionated heparin: Patients in the dilute heparin arm will receive a systemic loading dose of heparin of 15 units per kilogram of weight by rapid intravenous bolus. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started. Heparin will be delivered as a solution of 2 units/mL and the infusion will be prepared with 2,000 units of heparin in 1,000 mL of 0.9% NaCl and delivered intravenously proximal to the dialysis filter.
- Standard Concentrated Heparin: Arm A will receive standard concentrated heparin and will be delivered as an intravenous infusion proximal to the dialysis filter.
  Standard concentration unfractionated heparin: Patients in the standard heparin arm will receive a systemic loading dose of heparin of 15 units per kilogram of weight by rapid intravenous bolus. Then a maintenance rate of heparin of 7.5 U/Kg per hour will be started and delivered in a standard concentration intravenously proximal to the dialysis filter via a syringe. The concentration of heparin used will be 1,000 units of heparin per 1 mL of 0.9% NaCl.
Period: Overall Study
Arm/Group | Dilute Heparin | Standard Concentrated Heparin
Started | 4 | 8
Completed | 3 | 4
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 1
Not completed — CRRT stopped for head CT | 0 | 1
Not completed — Death | 0 | 1
Not completed — CRRT stopped for head MRI | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dilute Heparin | Standard Concentrated Heparin | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.25 (16.5) | 57.5 (11) | 57.75 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Filter Life
Description: The primary endpoint for this study will be the difference in filter life in hours between the group receiving dilute heparin and the group receiving standard concentrated heparin.
Time Frame: 72 hours
Population: analysis does not include those that had dialysis stopped before end of filter life
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dilute Heparin | Standard Concentrated Heparin
Number analyzed (Participants) | 3 | 4
hours | 22.46 (3.32) | 33 (22.22)

2. Secondary Outcome: Number of Major Bleeding Complications
Description: Information on major bleeding complications, and need for blood product transfusions will be collected.
Time Frame: 72 hours
Population: includes all that started study
Measure: Number; unit: clinical active major bleeding episodes
Arm/Group | Dilute Heparin | Standard Concentrated Heparin
Number analyzed (Participants) | 4 | 8
clinical active major bleeding episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: 72 hours from start of dialysis
Arm/Group | Dilute Heparin | Standard Concentrated Heparin
All-Cause Mortality (participants affected / at risk) | 2/4 | 4/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No